CLINICAL TRIAL: NCT03406988
Title: Regional Grafting of Autologous Adipose Tissue in the Treatment of Systemic Sclerosis Digital Ulcers: a Prospective Randomized Controlled Study
Brief Title: Autologous Adipose Tissue in the Treatment of Systemic Sclerosis Digital Ulcers
Acronym: ADUL-SSc
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ASST Gaetano Pini-CTO (Other)
Collaborators: Società Italiana di Reumatologia (Unknown)
Responsible Party: Principal Investigator, Nicoletta Del Papa, MD, Head of the Scleroderma Clinics, Rheumatology Department, ASST Gaetano Pini-CTO
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ID Sperimentazione 138
Record Dates: First submitted 2018-01-08; First posted 2018-01-23 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Systemic Sclerosis; Digital Ulcer
Keywords: Systemic Sclerosis; Digital Ulcer; Autologous fat grafting; Adipose tissue stem cells
MeSH Terms: conditions — Scleroderma, Systemic; digital ulcers | interventions — Nifedipine

STUDY DESIGN:
Intervention Model Description: Candidate SSc patients will have only one active DU of at least 6 mm in diameter, lasting for at least 6 weeks, despite conventional vascular therapy. Patients with severe visceral manifestations, diabetes and treated with immune-suppressors and endothelin inhibitors will be excluded. Active therapy: implantation of 0.5-1 ml of autologous AT at the base of the finger with DU. Autologous AT will be obtained by liposuction from abdominal fat.
  SP will be blindly performed in the control group to simulate the AT-G. A false liposuction will be performed followed by the injection of 0.5-1 ml of 0.9% saline solution at the base of the affected finger. Basal therapy: weekly iloprost infusion (0.5-2 ng/Kg/min), and calcium-channel blockers (oral nifedipine 20 mg daily) will be continued during the entire observation time in all of the patients recruited in both arms of the study. The administration of analgesics to alleviate the DU-related pain will be also allowed for each patient.
Who Masked: Participant, Outcomes Assessor
Masking Description: Each enrolled patient will be blind regarding the administered therapy (active and sham procedure).
  Evaluation of primary and secondary outcomes will be performed by assessors blind regarding the administered therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autologous fat grafting (Experimental): Implantation of 0.5-1 ml of autologous AT at the base of the finger with DU.
  Interventions: Procedure: Autologous fat grafting
- Sham procedure (Placebo Comparator): False liposuction followed by the injection of 0.5-1 ml of 0.9% saline solution at the base of the affected finger.
  Interventions: Procedure: Sham procedure

INTERVENTIONS:
Procedure: Autologous fat grafting — Implantation of small amount of autologous adipose tissue at the base of the finger to induce a rapid healing of the distally located DU
  Other Names: Iloprost infusion, oral nifedipine
  Arms: Autologous fat grafting
Procedure: Sham procedure — Local injection of 0.5ml saline solution after a simulated liposuction procedure.
  Other Names: Iloprost infusion, oral nifedipine
  Arms: Sham procedure

SUMMARY:
A randomized controlled trial will be performed to confirm preliminary uncontrolled data indicating that regional adipose tissue grafting is effective in inducing digital ulcer healing in patients with systemic sclerosis.

Systemic Sclerosis patients with digital ulcers will be randomized to be blindly treated with adipose tissue implantation or a sham procedure. Adipose tissue grafting will consist of injection at the base of the finger with digital ulcer of 0.5-1 ml of adipose tissue after centrifugation of fat aspirate. Sharm procedure will consist of false liposuction and local injection of saline solution.

The primary end-point will be to compare the cumulative prevalence of healed digital ulcers in the two groups within the following 8 weeks.

DETAILED DESCRIPTION:
Systemic sclerosis (SSc) is an autoimmune disease characterized by a multifactorial pathological process where a central role is played by the progressive loss of the microvascular bed, with the consequent fibrotic changes in the involved organs and tissues.

The most advanced stages of capillary loss may induce the formation of digital ulcers (DUs) on the fingertips.The healing of DUs is often a lengthy process requiring accurate and intensive topical and systemic treatment. Nevertheless, in a significant number of cases this therapeutic approach is ineffective and distal necrosis with subsequent tissue loss or phalangeal amputation may eventually occur.

In a recent open pilot study performed by Del Papa et al., it has been demonstrated that autologous adipose tissue grafting (AT-G), which is known to contain both adipose-derived stem cells and a stromal/vascular fraction, was effective in inducing prompt healing of long lasting DUs localized in the fingertips of a small number of patients with SSc. The DU healing was accompanied by the rapid disappearance of local ischemic pain and evidence of a partial restoration of the capillary bed in the digits when assessed by nailfold videocapillaroscopy (NVC).

With the purpose of confirming these preliminary results, the investigators have designed a monocentric randomized controlled study. In accordance with the study protocol, patients with a typical SSc-related DU on the fingertip will be randomized to undergo a regional AT-G with autologous fat as active therapy or a 'sham' procedure (SP) - that simulates the active treatment - as placebo treatment. All of the patients with SSc enrolled in both arms will be blind regarding the treatment received. Furthermore, during the study period all of the enrolled patients will receive the same systemic vasoactive and topical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients candidate for enrollment in the study have to meet the 2013 classification criteria of the American College of Rheumatology/European League Against Rheumatism for SSc;
* Patients may have either the limited cutaneous or the diffuse cutaneous variants of SSc;
* All of the candidate patients must have only one active DU (cardinal ulcer), lasting for at least 6 weeks prior to enrolment time and showing no tendency to heal despite intravenous iloprost (0.5-2 ng/Kg/min), the oral administration of calcium-channel blockers (nifedipine) and local medication with surgical removal of necrotic tissue.

Exclusion Criteria:

* Presence of severe extra-cutaneous manifestations, such as cardiac, lung and renal involvement;
* Concomitant treatment with immune-suppressive therapies (including prednisone equivalent >10 mg);
* Current therapy with dual and selective endothelin inhibitors;
* Concomitant diabetes and/or other vascular diseases;
* Current pregnancy or breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2017-07-18 (Actual); Primary Completion 2018-03-31 (Estimated); Study Completion 2018-03-31 (Estimated)

PRIMARY OUTCOMES:
Digital Ulcer healing | 8 weeks after either autologus fat grafting or sham procedure.
  Prevalence of DU healing in the arm treated with autologous fat grafting in comparison with the prevalence of healing in the placebo group.

SECONDARY OUTCOMES:
Pain evaluation by Visual Analogue Scale (VAS) | This evaluation will be done at baseline and at the 2nd, 4th, 6th, 8th week after interventions (either autologus fat grafting or sham procedure).
  The pain VAS is a continuous scale comprised of a horizontal line of 10 centimeters (100 mm) in length, ranging from 0 (minimum= no pain) to 100 (worst imaginable pain). The respondents will be asked to place a line perpendicular to the VAS line at the point that represents their pain intensity. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100.
  In this study VAS score will be used to measure the decrease (or resolution) of pain with respect to baseline value in patients who will undergo treatment with autologous fat grafting (active arm) in comparison with patients of the placebo group.
Neovascularization evaluation | Baseline and 8 weeks after either autologus fat grafting or sham procedure.
  Increase of the number of capillaries assessed by NVC in the affected digit of patients treated with autologous fat grafting in comparison with patients of the placebo group.

CONTACTS AND LOCATIONS:
Overall Officials: Nicoletta Del Papa, MD, Principal Investigator — ASST Gaetano Pini-CTO
Locations (1):
- UOC Day Hospital Reumatologia, ASST G. Pini-CTO, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gabrielli A, Avvedimento EV, Krieg T. Scleroderma. N Engl J Med. 2009 May 7;360(19):1989-2003. doi: 10.1056/NEJMra0806188. No abstract available. PMID 19420368
- [Background] Steen V, Denton CP, Pope JE, Matucci-Cerinic M. Digital ulcers: overt vascular disease in systemic sclerosis. Rheumatology (Oxford). 2009 Jun;48 Suppl 3:iii19-24. doi: 10.1093/rheumatology/kep105. PMID 19487218
- [Background] Del Papa N, Di Luca G, Sambataro D, Zaccara E, Maglione W, Gabrielli A, Fraticelli P, Moroncini G, Beretta L, Santaniello A, Sambataro G, Ferraresi R, Vitali C. Regional implantation of autologous adipose tissue-derived cells induces a prompt healing of long-lasting indolent digital ulcers in patients with systemic sclerosis. Cell Transplant. 2015;24(11):2297-305. doi: 10.3727/096368914X685636. Epub 2014 Dec 12. PMID 25506730
- [Derived] Del Papa N, Di Luca G, Andracco R, Zaccara E, Maglione W, Pignataro F, Minniti A, Vitali C. Regional grafting of autologous adipose tissue is effective in inducing prompt healing of indolent digital ulcers in patients with systemic sclerosis: results of a monocentric randomized controlled study. Arthritis Res Ther. 2019 Jan 7;21(1):7. doi: 10.1186/s13075-018-1792-8. PMID 30616671